CLINICAL TRIAL: NCT05353842
Title: Scale Up Trial of Project WOWii to Increase Exercise Among People With Spinal Cord Injury (SCI)
Brief Title: Scale Up of Project Workout on Wheels Internet Intervention (WOWii)
Acronym: WOWii
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: Kessler Institute for Rehabilitation (Industry); Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Katherine Froehlich-Grobe, Research Scientist, Craig Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 901FRE0046-01-01
Record Dates: First submitted 2022-01-03; First posted 2022-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WOWii Intervention (Experimental): Workout on Wheels Internet Intervention (WOWii) program which includes: 1) WOWii website to guide participants in an exercise program, 2) home exercise starter program; 3) weekly support from a peer facilitator via online (video) meetings.
  Interventions: Behavioral: WOWii Program

INTERVENTIONS:
Behavioral: WOWii Program — Workout on Wheels Internet Internvention (WOWii) which includes: 1) WOWii website to guide participants in an exercise program, 2) home exercise starter program; 3) weekly support from a peer facilitator via online (video) meetings.

SUMMARY:
This study is designed is to test the feasibility, fidelity, and effectiveness of scaling up an evidence- and theory-based virtually delivered physical activity intervention (WOWii) for individuals living with chronic SCI for delivery through other rehabilitation settings. The study outcomes address (1) feasibility based on participant enrollment, retention, and program engagement; (2) fidelity of intervention delivery; and (3) program effectiveness based on subjective and objective exercise data, and participant exercise perceptions regarding self-efficacy and barriers.

ELIGIBILITY:
Inclusion Criteria:

* more than 12 months post SCI
* requires use of wheelchair due to SCI
* receive signed approval from medical provider to initiate moderate-intensity exercise program
* have internet access via computer, tablet, or smartphone
* provide informed consent

Exclusion Criteria:

* already engaged in engaged in sufficient physical activity to meet CDCP guidelines
* cognitive of language impairments that would affect ability to participate
* presence of medical issue for which exercise is contraindicated
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment of Participants in WOWii Program (feasibility) | One time at end of study recruitment
  Total number of participants enrolled at each site
Retention of Participants Enrolled in WOWii Program (feasibility) | One time at end of 16 week intervention
  Total number of WOWii sessions attended
Engagement of Participants Enrolled in WOWii Program (feasibilty) | One time at end of 16 week intervention
  Total number of WOWii online activities completed
Percentage of behavior skills covered by peer facilitators during WOWii Program (fidelity) | One time at end of 16 week intervention
  Percentage of items on fidelity check list that are marked as completed
% of WOWii sessions in which peer facilitators generate group-based conversation (fidelity) | One time at end of 16 week intervention
  % of sessions on fidelity check list that are marked as having grop-based conversation
Change in number of minutes spent in aerobic exercise (effectiveness) | Baseline, end of intervention (Week 16), end of follow up (Week 24)
  Objective measure of change in activity level
Change in score on International Physical Activity Questionnaire Scores (effectiveness) | Baseline, end of intervention (Week 16), end of follow up (Week 24)
  8-item survey asking days/week and minutes/day spent in various physical activities.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Shepherd Center, Atlanta, Georgia
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: No